CLINICAL TRIAL: NCT05494008
Title: Evaluation of Effectiveness and Safety of Korean Herbal Medicine Treatment Strategy for Outpatients With Post-accident Syndromes After Acute Phase: A Pilot Pragmatic Randomized Controlled Trial
Brief Title: Evaluation of Effectiveness and Safety of Korean Herbal Medicine for Post-accident Syndromes After Acute Phase
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Principal Investigator, In-Hyuk Ha, KMD, Director, Jaseng Medical Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JS-CT-2021-09
Record Dates: First submitted 2022-08-05; First posted 2022-08-09 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Traffic Accident; Whiplash Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Korean herbal medicine treatment (Experimental): The Korean herbal medicine treatment group received Korean herbal medicine treatment for 28 days. A trained doctor of Korean medicine with at least 3 years of clinical experience prescribed Korean herbal medicine.
  The Korean herbal medicine treatment group were also treated with other Korean medical treatment for twice a week for 4 weeks: acupuncture, pharmacoacupuncture, cupping, and chuna.
  Interventions: Procedure: Korean herbal medicine treatment
- Non-Korean herbal medicine treatment (Active Comparator): The control group received Korean medical treatment for twice a week for 4 weeks: acupuncture, pharmacoacupuncture, cupping and chuna. (except Korean herbal medicine)
  Interventions: Procedure: Non-Korean herbal medicine treatment

INTERVENTIONS:
Procedure: Korean herbal medicine treatment — Korean herbal medicine treatment is a treatment using complex extract of medicinal herbs prescribed by a Korean medicine doctor who has completed specialized education to diagnose the health condition and symptoms of patients with post-traffic accident syndromes.
  Arms: Korean herbal medicine treatment
Procedure: Non-Korean herbal medicine treatment — acupuncture, pharmacoacupuncture, cupping, chuna
  Arms: Non-Korean herbal medicine treatment

SUMMARY:
This study is a single blind, randomized controlled trail. condition/disease: Post-accident syndromes after acute phase treatment/intervention: herbal medicine treatment strategy

DETAILED DESCRIPTION:
The Korean herbal medicine is a complex extract of medicinal herbs prescribed by a Korean medicine doctor who has completed specialized education to diagnose the health condition and symptoms of patients with post-traffic accident syndromes. This treatment is known to relieve the post-accident syndromes and improve health. However, there are no studies examining the efficacy of Korean herbal medicine alone.

So, the investigators will conduct a randomized controlled trials to verify the efficacy and safety of Korean herbal medicine. From July, 2021 to May, 2022, the investigators recruited 40 patients who are suffered from post-accident syndromes with the numeric rating scale(NRS) over 5. For experimental group(the Korean herbal medicine treatment group, n=20), the investigators conducted Korean medicine treatment for 4 weeks(28 days), and for control group(the Non-Korean herbal medicine treatment group, n=20), just Korean medical treatment(acupuncture, pharmacoacupuncture, cupping, and chuna) has been conducted. For these two groups, the investigators compared NRS, Impact of Event Scale-Revised-Korean(IES-R-K), 5-level EuroQol 5-dimension(EQ-5D-5L), Short-Form-12 Health Survey version2(SF-12 v2), and Patient Global Impression of Change(PGIC).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19-70 years on the date they sign the consent form
* Patients who have passed more than 8 weeks but less than 24 weeks from the date of the accident on the date they sign the consent form
* Patients with NRS ≥ 5 for post-accident syndromes
* Patients who provide consent to participate in the trial and return the informed consent form

Exclusion Criteria:

* Patients whose pain is not due to a traffic accident but due to an existing disease (hernia of intervertebral discs, spinal canal stenosis, fibromyalgia, etc.)
* Patients who have undergone surgery due to the current traffic accident
* Patients with progressive neurological deficits or with severe neurological symptoms
* Patients with other chronic conditions that may interfere with the interpretation of the therapeutic effects or results: cardiovascular disease, kidney disease, diabetic neuropathy, dementia, epilepsy, etc.
* Patients who are taking steroids, immunosuppressants, mental illness drugs, or other drugs that may affect the results of the study
* Patients with exceeding twice the normal value in liver function tests and kidney function tests in screening tests
* Patients with kidney or liver/biliary system disease (hepatitis, fatty liver, cirrhosis, liver cancer, biliary obstruction, etc.)
* Patients with gastrointestinal dysfunction or patients who have had a surgery that may affect drug absorption, such as gastrectomy
* Patients who are pregnant or planning to become pregnant
* Patients with a serious mental illness
* Patients who are participated in clinical trials other than observational studies without therapeutic intervention.
* Patients who are difficult to complete the research participation agreement
* Other patients whose participation in the trial is judged by a researcher to be problematic

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-07-24 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-09-13 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale(NRS) of post-accident syndromes | Change from baseline to 4 months
  The severity of post-accident syndrome will be assessed using NRS. NRS is a scale in which the patient indicates their subjective severity of symptoms as a whole number from 0 to 10. The participant is asked to report their severity of post-accident syndrome using NRS, where 0 indicates 'no pain or discomfort' and 10 indicates 'the most severe pain and discomfort imaginable'.

SECONDARY OUTCOMES:
Numeric Rating Scale(NRS) of musculoskeletal complaints of post-accident syndromes | Baseline(week 1-1), week 3-1, week 5, week 9, week 17
  The severity of musculoskeletal complaints of post-accident syndrome will be assessed using NRS. The participant is asked to report their severity of musculoskeletal complaints(post neck pain, lower back pain, shoulder pain, knee pain, etc) using NRS, where 0 indicates 'no pain or discomfort' and 10 indicates 'the most severe pain or discomfort imaginable'.
Numeric Rating Scale(NRS) of neurological complaints of post-accident syndromes | Baseline(week 1-1), week 3-1, week 5, week 9, week 17
  The severity of neurological complaints of post-accident syndrome will be assessed using NRS. The participant is asked to report their severity of neurological complaints(headache, dizziness, etc) using NRS, where 0 indicates 'no discomfort' and 10 indicates 'the most severe discomfort imaginable'.
Numeric Rating Scale(NRS) of psychiatric complaints of post-accident syndromes | Baseline(week 1-1), week 3-1, week 5, week 9, week 17
  The severity of psychiatric complaints of post-accident syndrome will be assessed using NRS. The participant is asked to report their severity of psychiatric complaints(anxiety, depression, anger, insomnia etc) using NRS, where 0 indicates 'no discomfort' and 10 indicates 'the most severe discomfort imaginable'.
Numeric Rating Scale(NRS) of digestive systemic complaints of post-accident syndromes | Baseline(week 1-1), week 3-1, week 5, week 9, week 17
  The severity of digestive systemic complaints of post-accident syndrome will be assessed using NRS. The participant is asked to report their severity of digestive systemic complaints(indigestion, loss of appetite, etc) using NRS, where 0 indicates 'no discomfort' and 10 indicates 'the most severe discomfort imaginable'.
Numeric Rating Scale(NRS) of general symptoms of post-accident syndromes | Baseline(week 1-1), week 3-1, week 5, week 9, week 17
  The severity of general symptoms of post-accident syndrome will be assessed using NRS. The participant is asked to report their severity of general symptoms(fatigue, powerlessness, etc) using NRS, where 0 indicates 'no discomfort' and 10 indicates 'the most severe discomfort imaginable'.
Impact of Event Scale-Revised-Korean (IES-R-K) | Baseline(week 1-1), week 3-1, week 5, week 9, week 17
  The IES-R-K is a 22-item self-report scale that evaluates subjective stress caused by traumatic events. Each item is rated on a scale of 0 (not at all) to 4 (extremely) of the severity of symptoms based on the past week, with a total score ranging from 0 to 88. Although it is not generally recommended for the diagnosis of PTSD, it is an evaluation scale widely used in trauma-related clinical studies.
5-level EuroQol 5-dimension (EQ-5D-5L) | Baseline(week 1-1), week 3-1, week 5, week 9, week 17
  The EQ-5D is a method of indirectly calculating the weights of certain health states for quality of life after a multidimensional investigation of health states, and is the most widely used instrument for this purpose. The EQ-5D consists of 5 questions about current health state (mobility, self-care, usual activities, pain, anxiety/depression), and each question is scored on a 5-point Likert scale (1=no problems, 3=moderate problems, 5=severe problems). In this study, the investigators will use the Korean version of the EQ-5D, which has been demonstrated to be valid.
Short-Form-12 Health Survey version2 (SF-12 v2) | Baseline(week 1-1), week 3-1, week 5, week 9, week 17
  SF-12 version 2 is a questionnaire that evaluates health-related quality of life (HRQoL). It consists of 12 items in 8 areas (physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional and mental health).
Patient Global Impression of Change (PGIC) | week 5, week 9, week 17
  The PGIC is an index that assesses improvements in post-accident syndromes caused by traffic accident. Participants rate the improvement in post-accident syndromes after treatment on a 7-point Likert scale (1=Very much improved, 4=No change, 7=Very much worse)
Economic evaluation question | Through study completion, an average of 4 months
  In order to measure cost items, a questionnaire with questions measuring medical expenses, non-medical expenses, time costs, productivity loss costs, etc. is used.
Drug Consumption | Through study completion, an average of 4 months
  Check the type and dose of drugs taken during the study period every visit
Adverse events | Through study completion, an average of 4 months
  Check adverse events every visit

CONTACTS AND LOCATIONS:
Overall Officials: In-Hyuk Ha, PhD, Principal Investigator — Jaseng Medical Foundation
Locations (1):
- Jaseng Hospital of Korean Medicine, Seoul, Gangnam-Gu, South Korea

IPD SHARING:
Plan to Share IPD: No